CLINICAL TRIAL: NCT02429180
Title: Community-based Rehabilitation Training After Stroke: a Pilot Randomised Controlled Trial
Brief Title: Rehabilitation Training After Stroke
Acronym: ReTrain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: The Stroke Association, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRF192
Record Dates: First submitted 2015-04-16; First posted 2015-04-29 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rehabilitation training (Experimental): ReTrain: an exercise-based functional training programme comprising two phases: (1) weekly supervised sessions; (2) monthly drop-in sessions, plus home-based exercise in each phase.
  * Week 1: one-to-one consultations with trainer to introduce programme, assess individual's concerns and capabilities, introduce and negotiate initial goals
  * Weeks 2-11: bi-weekly 90 minute group class with group-based activities and one-to-one coaching, based on ongoing goal negotiation review and progression.
  * Week 12: one-to-one consultations with trainer to review goals and plan ongoing unsupervised exercise programme
  * Weeks 13-24: monthly drop-in sessions for one-to-one consultation, support and progression.
  Interventions: Other: Rehabilitation
- Control (No Intervention): Control: treatment as usual plus receipt of a UK Stroke Association booklet on exercise after stroke.

INTERVENTIONS:
Other: Rehabilitation — ReTrain: an exercise-based functional training programme comprising two phases: (1) weekly supervised sessions; (2) monthly drop-in sessions, plus home-based exercise in each phase.
  * Week 1: one-to-one consultations with trainer to introduce programme, assess individual's concerns and capabilities, introduce and negotiate initial goals
  * Weeks 2-11: bi-weekly 90 minute group class with group-based activities and one-to-one coaching, based on ongoing goal negotiation review and progression.
  * Week 12: one-to-one consultations with trainer to review goals and plan ongoing unsupervised exercise programme
  * Weeks 13-24: monthly drop-in sessions for one-to-one consultation, support and progression.
  Arms: Rehabilitation training

SUMMARY:
A pilot study that will evaluate the feasibility and acceptability of procedures to inform the design and delivery of a definitive RCT of ReTrain (which would assess the clinical and cost effectiveness of ReTrain for stroke survivors).

DETAILED DESCRIPTION:
Background and rationale

Residual physical disability is common following discharge from stroke rehabilitation services. A third of first-time stroke survivors remain physically disabled five years after their stroke, equivalent to more than 300,000 people in the UK. Stroke services are traditionally "front loaded" with provision tailing off a few months after stroke. However, people with stroke report a variety of unmet long-term needs and a sense of being abandoned by NHS services. The UK National Stroke Strategy recommends that stroke be regarded as a Long Term Condition and that continuing support is provided for those who need it. This includes community-based rehabilitation, with an emphasis on personalisation, re-ablement and self-management of the consequences of stroke. There is good evidence that exercise can promote functional recovery, enhance adjustment and coping, improve psychological wellbeing, and reduce the risk of recurrence. Hence stroke guidelines recommend that people with stroke should regularly engage in specific forms of exercise, however many do not meet these recommendations. Various personal and environmental factors may account for this: stroke-related impairments, lack of confidence or knowledge regarding exercise and its benefits, and inadequate provision of support programmes and facilities. In response, community-based programmes are being offered. However, these programmes often focus on fitness rather than function, giving little attention to self-management or to sustaining behaviour (to ensure benefits are maintained after structured programmes have ended). National stroke guidelines recommend interventions address functional improvement and self-management strategies even though a recently updated Cochrane review notes the gap in evidence regarding these interventions.

An approach called ARNI (Action for Rehabilitation from Neurological Injury) attempts to address these concerns; it was created specifically for people with stroke and acquired brain injury who wish to continue their functional recovery.ARNI is not a rigidly-defined programme but a set of principles and strategies tailored to individual circumstances and contexts. It is led by registered exercise professionals who have been additionally trained and accredited by the ARNI institute (http://www.arni.uk.com). In the UK, the NHS, Local Authorities and other organisations are using ARNI trainers to provide community-based training for stroke survivors. Our survey of this training included Northeast England, Lancashire, Luton and Bedfordshire, Milton Keynes, Hillingdon and Cornwall. The survey found that training has been very positively received by stroke survivors, their families and clinicians but it varied in content and delivery. Reports of benefits by the broadcaster Andrew Marr have also increased public awareness of ARNI. However the evidence for ARNI remains largely anecdotal, it may only work for a selected few and the approach is difficult to replicate. There is a need for a more detailed cohesive specification of ARNI that could be rigorously evaluated and replicated. Furthermore a stroke survivor participating in our Institution's research question generation process asked if ARNI worked but as yet there have been no randomised controlled trials (RCTs) of this intervention. Thus we have followed the Medical Research Council's framework for the development and evaluation of complex interventions and undertaken five linked preliminary studies: 1) a survey of current ARNI provision in the UK; 2) a comparison of the ARNI approach with relevant stroke practice guidelines, 3) before-and-after studies of both group-based and 4) one-to-one training and 5) focus groups conducted with our participants. From this work we have designed a programme called ReTrain (Rehabilitation Training) which is based on core ARNI principles and informed by best practice guidelines for stroke. Before undertaking a large definitive RCT of ReTrain a pilot study is needed to address issues of feasibility and acceptability.

Purpose of the study

ReTrain aims to improve (i) functional mobility, (ii) adherence to national guidelines on post-stroke exercise levels, and (iii) health-related quality of life, for people after stroke who have been discharged from clinical rehabilitation. A definitive RCT is required to assess the clinical and cost effectiveness of the ReTrain intervention. The purpose of this pilot study is to assess to feasibility of such a trial and to evaluate trial procedures to inform the design of a definitive trial.

ELIGIBILITY:
Inclusion Criteria:

* Primary clinical diagnosis of stroke (assessed by referring clinician/GP records)
* >1 month (but no upper limit) since discharge from NHS physical rehabilitation services at randomisation
* Able to walk independently indoors with or without mobility aids, but has self-reported difficulty or requires help on stairs, slopes or uneven surfaces (assessed by recruiting team using standard tools)
* Willingness to be randomised to either control or ReTrain (and attend the training venue)
* Cognitive capacity and communication ability sufficient to participate in the study (assessed by recruiting team using standard tools).24 NB: Criterion (3) has been selected pragmatically to maximise eligibility while ensuring participants have a mobility deficit that could be addressed by the intervention. Eligible people with aphasia will not be excluded.

Exclusion Criteria:

* <18 years old
* Contraindications to moderate to vigorous physical activity. Used in GP screening assessment form. (Adapted from ACSM guidelines 25) Contraindications include:

  * Acute or uncontrolled heart failure
  * Unstable or uncontrolled angina
  * Uncontrolled cardiac dysrhythmia causing symptoms or haemodynamic compromise
  * Symptomatic severe aortic stenosis
  * Current deep vein thrombosis, pulmonary embolus or pulmonary infarction
  * Acute myocarditis or pericarditis
  * Suspected or known dissecting aneurysm
  * Unstable / uncontrolled blood pressure
  * Systolic blood pressure > 160
  * Diastolic blood pressure > 100
  * Acute systemic infection
  * Uncontrolled diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2015-07-31 (Actual); Primary Completion 2016-01-27 (Actual); Study Completion 2016-01-27 (Actual)

PRIMARY OUTCOMES:
Change in Rivermead Mobility index | Baseline, 6 months, 9 months
  15-item, dichotomously scored measure of mobility disability. Fourteen items are self-report and one (standing for 10s without aids) is scored by observation
Change in Timed Up and Go Test | Baseline, 6 months, 9 months
  Objective measure of mobility, balance and locomotor performance, in which the individual is observed and timed rising from a chair, walking 3m, turning and returning to the chair
Change in Modified Patient Specific Functional Scale | Baseline, 6 months, 9 months
  Identification by individual of up to five functional tasks that are important and difficult to perform, and rating of ability to perform each task on a 0-10 scale
Change in Physical Activity Diary | Baseline, 6 months, 9 months
  Participants record the type of activity and its duration each day of the week (1-2 minutes per day to complete).
Change in Physical activity - 7-day accelerometry | Baseline, 6 months, 9 months
  Worn by individual to assess physical activity behaviour over seven days. Should take 5 minutes to fit watch and 10 minutes to post back

SECONDARY OUTCOMES:
Fatigue Assessment Scale | Baseline, 6 months, 9 months
  10-item self-completion questionnaire in which aspects of fatigue are rated on how regularly they are experienced, using a 5-point scale
Stroke Self-efficacy Questionnaire | Baseline, 9 months
  10-item questionnaire in which participants rate their confidence in completing some tasks that may have been difficult for them since their stroke
Exercise beliefs questionnaire | Baseline, 9 months
  Measures attitudes to exercise by rating levels of agreement to 5 statements about what it can achieve for the individual.
Exercise self-efficacy questionnaire | Baseline, 9 months
  Self-rating of confidence to overcome 4 personal barriers to exercise
Stroke Quality of Life | Baseline, 9 months
  Self-rating of twelve dimensions of lifestyle and personal functioning
EQ-5D-5L | Baseline, 9 months
  Measuring health-related quality of life and can be used for cost utility analysis
SF-12 46 | Baseline, 9 months
  Abbreviated version of the Short-Form-36 self-completion questionnaire measuring health-related quality of life. It can also be used to calculate the SF-6D, which may be used for cost utility analysis.
Service Receipt Inventory | Baseline, 9 months
  Record of types and amount of use of health and social care resources including medication, clinical contacts, formal and informal social care. Completed by Assessor drawing on participant and family accounts, and clinical records if available.
Carer Burden Index | Baseline, 9 months
  Carers of stroke survivors rate the difficulties and challenges of providing care
Adverse incidents | 6 months, 9 months
  Adverse events

OTHER OUTCOMES:
The type and frequency of health and allied services measured using an adapted Client Service Receipt Inventory based on the TRACS study | 0-9 months
  Collection of service use data

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Dean, PhD, Study Chair — University of Exeter Medical School; Rod Taylor, Prof, Study Director — University of Exeter Medical School; Anne Forster, Prof, Study Director — University of Leeds; Anne Spencer, Prof, Study Director — University of Exeter Medical School; Martin James, Dr, Study Director — Royal Devon and Exeter NHS Foundation Trust; Rhoda Allison, Dr, Study Director — Torbay & Southern Devon Health & Care Trust; Shirley Stevens, Mrs, Study Director — PenPIG; Meriel Norris, Dr, Study Director — Brunel University; Leon Poltawski, Dr, Study Director — University of Exeter Medical School
Locations (1):
- University of Exeter Medical School, Exeter, Devon, United Kingdom

REFERENCES:
- [Derived] Taylor E, Soilemezi D, Urquhart DS, Cunningham S, Lewis S, Neilson AR, Ensor H, Vogiatizis I, Allen L, Saynor ZL; ExACT-CF study group. Exploring Exercise as Airway Clearance in Cystic Fibrosis: A Qualitative Study From the ExACT-CF Feasibility Trial. Pediatr Pulmonol. 2026 Jan;61(1):e71470. doi: 10.1002/ppul.71470. PMID 41587390
- [Derived] Hollands L, Calitri R, Warmoth K, Shepherd A, Allison R, Dean S; ReTrain Trial; team. Assessing the fidelity of the independently getting up off the floor (IGO) technique as part of the ReTrain pilot feasibility randomised controlled trial for stroke survivors. Disabil Rehabil. 2022 Dec;44(25):7829-7838. doi: 10.1080/09638288.2021.1998672. Epub 2021 Nov 12. PMID 34767488
- [Derived] Norris M, Poltawski L, Calitri R, Shepherd AI, Dean SG; ReTrain Team. Hope and despair: a qualitative exploration of the experiences and impact of trial processes in a rehabilitation trial. Trials. 2019 Aug 23;20(1):525. doi: 10.1186/s13063-019-3633-8. PMID 31443735
- [Derived] Norris M, Poltawski L, Calitri R, Shepherd AI, Dean SG; ReTrain Team. Acceptability and experience of a functional training programme (ReTrain) in community-dwelling stroke survivors in South West England: a qualitative study. BMJ Open. 2018 Jul 25;8(7):e022175. doi: 10.1136/bmjopen-2018-022175. PMID 30049699
- [Derived] Dean SG, Poltawski L, Forster A, Taylor RS, Spencer A, James M, Allison R, Stevens S, Norris M, Shepherd AI, Landa P, Pulsford RM, Hollands L, Calitri R. Community-based rehabilitation training after stroke: results of a pilot randomised controlled trial (ReTrain) investigating acceptability and feasibility. BMJ Open. 2018 Feb 15;8(2):e018409. doi: 10.1136/bmjopen-2017-018409. PMID 29449290
- [Derived] Dean SG, Poltawski L, Forster A, Taylor RS, Spencer A, James M, Allison R, Stevens S, Norris M, Shepherd AI, Calitri R. Community-based Rehabilitation Training after stroke: protocol of a pilot randomised controlled trial (ReTrain). BMJ Open. 2016 Oct 3;6(10):e012375. doi: 10.1136/bmjopen-2016-012375. PMID 27697876
- See also: Action for rehabilitation after neurological injury — http://www.arni.uk.com/
- See also: PenCLAHRC — http://clahrc-peninsula.nihr.ac.uk/